CLINICAL TRIAL: NCT07125976
Title: The Effect of Peer Support on Disease Adaptation and Self-Care Ability in Individuals Diagnosed With Chronic Kidney Failure
Acronym: Peer support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: pınar dogan (Other)
Responsible Party: Sponsor-Investigator, pınar dogan, Asst.Prof., Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 29384756
Record Dates: First submitted 2025-07-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: Chronic Kidney Disease; Disease Adaptation; Self-care Ability; Peer Interaction
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Experimental study with pre-post test control group
Who Masked: Participant
Masking Description: patients with chronic kidney disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Support group (Experimental): In this group, structured peer support was provided for 1 week in addition to routine care practices applied in the clinic.
  Interventions: Behavioral: peer support
- Control group (No Intervention): group monitored with routine clinical care

INTERVENTIONS:
Behavioral: peer support — This intervention is a one-week, structured peer support program for patients in the first six months of hemodialysis treatment.
  Arms: Peer Support group

SUMMARY:
This study was designed as an interventional, pretest-posttest controlled trial to examine the effects of peer interaction on disease adaptation and self-care ability in patients newly diagnosed with chronic kidney failure and starting dialysis. The main hypothesis:

H1: Structured peer support provided to patients receiving hemodialysis treatment has a positive effect on their level of adaptation to the disease.

H2: Structured peer support provided to patients receiving hemodialysis treatment has a positive effect on their self-care power.

Researchers will compare control group to see if adaptation to the dieases and self-care power.

Patients in the intervention group received peer support during their hospital stay, while those in the control group followed the routine clinical process.

DETAILED DESCRIPTION:
This study was conducted with 64 patients in the nephrology clinic of a Training and Research Hospital in Istanbul. Data were collected using the Personal Information Form, the Chronic Illness Adaptation Scale, and the Self-Management of Chronic Illness Scale. Patients in the intervention group received peer support during their hospital stay, while those in the control group followed the routine clinical process. Participants in the intervention group took part in a structured peer support program, with pre-test data collected through the Self-Care Management Scale in Chronic Illness and the Chronic Illness Adaptation Scale. The program consisted of 4-6 sessions over one week, each lasting 30-45 minutes, focusing on disease information, self-care behaviors, psychosocial coping, and motivation, delivered by trained peers of similar age and gender. Post-test data were collected after the program to assess changes and analyze the effect of structured peer support.

ELIGIBILITY:
Inclusion Criteria:

* Those receiving hemodialysis treatment for at most 6 months
* Not having mental illness according to DSM
* Without multiple chronic diseases
* Who agreed to participate in the study

Exclusion Criteria:

* Hospital stay longer or shorter than 1 week
* Treatment complications developed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Chronic disease adaptation scale | Day 1, upon hospital admission) and at discharge (average of 7 days after admission.
  It was used to determine the level of adaptation of hemodialysis patients to the disease. The minimum possible score on the scale is 25, and the maximum is 125. Higher scores on the scale indicate an increased level of adaptation to the illness.
Self-care management scale | Day 1, upon hospital admission) and at discharge (average of 7 days after admission.
  It was used to measure patients' ability to manage their self-care. The possible score on the scale ranges from 35 to 175, and higher scores indicate better self-care management.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protokol may be share for 1 year
Supporting Information: Study Protocol
Time Frame: It can be shared for 1 year after September 1, 2025.